CLINICAL TRIAL: NCT06717607
Title: Comparing Visual Outcomes in Matched Patients Receiving a Low Cylinder Power Toric IOL or a Non-toric IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ifocus Oyeklinikk (Network)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Morten Gundersen, MD, Ifocus Oyeklinikk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGG-2021-01; 370677 (Other: REK Norway Ethics Committee)
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Cataract and IOL Surgery
Keywords: Toric IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Clareon T2 IOL implantation (Experimental): low cylinder toric IOL
  Interventions: Device: low cylinder toric IOL
- Clareon non-toric IOL implantation (Active Comparator): Non-toric IOL
  Interventions: Device: non-toric IOL implantation

INTERVENTIONS:
Device: low cylinder toric IOL — Clareon T2 toric IOL implantation
  Other Names: Clareon T2 IOL implantation
  Arms: Clareon T2 IOL implantation
Device: non-toric IOL implantation — Clareon non-toric IOL
  Other Names: Clareon non-toric IOL implantation
  Arms: Clareon non-toric IOL implantation

SUMMARY:
The purpose of the study is to determine if visual function is improved with implantation of a low-cylinder toric intraocular lens, relative to a non-toric intraocular lens.

DETAILED DESCRIPTION:
The Clareon(R) T2 IOL and the Clareon (R) non-toric IOL will be randomly implanted in subjects determined to be appropriate for the T2 IOL. Visual acuity, low contrast acuity and contrast sensitivity will be measured 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* candidate for cataract surgery, suitable for implantation with a low cylinder toric IOL

Exclusion Criteria:

* pathology that would confound outcomes, previous ocular surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity (UDVA) | 3 months
  UDVA (logMAR)

SECONDARY OUTCOMES:
Mean refraction, spherical equivalent (MRSE) | 3 months
  MRSE, diopters
Manifest refractive cylinder | 3 months
  Manifest cylinder, diopters
Percentage of eyes with <= 0.25 D of refractive cylinder | 3 months
  As above
Percentage of eyes with <= 0.50 D of refractive cylinder | 3 months
  As above
Corrected distance visual acuity | 3 months
  CDVA, logMAR
Mesopic contrast sensitivity | 3 months
  Contrast sensitivity curve
Photopic contrast sensitivity | 3 months
  Contrast sensitivity curve
Low contrast visual acuity | 3 months
  Visual acuity (VA), logMAR

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Gunnar Gundersen, MD, PhD, Principal Investigator — Ifocus Oyeklinikk
Locations (1):
- Ifocus øyeklinikk, Haugesund, Norway

DOCUMENTS (1):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT06717607/Prot_000.pdf